CLINICAL TRIAL: NCT02388100
Title: The Glycemia Reduction Approaches in Diabetes: a Comparative Effectiveness Study (GRADE Study) Capillary Blood Collection: a Pilot Study
Brief Title: The GRADE Capillary Blood Collection Pilot Study
Status: Completed | Type: Observational
Sponsor: GRADE Study Group (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: GRADE_CAP; 1U01DK098246-01 (NIH)
Record Dates: First submitted 2015-03-06; First posted 2015-03-13 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Capillary HbA1c collection

SUMMARY:
This pilot study is planned to validate the comparability of HbA1c results obtained from whole blood collection via venous phlebotomy versus a capillary collection of whole blood. The participant will self-collect capillary blood into HbA1c prep vials containing a buffer; these prep vials will be sent to the CBL at ambient temperature via US Postal System (USPS) mail. The feasibility of self-collection of these capillary samples by GRADE participants will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Current GRADE participant with a scheduled follow-up visit

Exclusion Criteria:

* GRADE participants attending first quarterly (Month 3) visit or an annual visit

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All GRADE study participants scheduled for a follow-up visit at selected GRADE clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
HbA1c obtained from venous versus capillary measurements at one point in time for each participant. | Cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: David Nathan, MD, Study Chair — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Southwestern American Indian Center, Phoenix, Arizona
  - University of Colorado, Denver, Colorado
  - Pacific Health Research and Education Institute (VA Pacific Islands), Honolulu, Hawaii
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - International Diabetes Center, Minneapolis, Minnesota

REFERENCES:
- [Background] Nathan DM, Krause-Steinrauf H, Braffett BH, Arends VL, Younes N, McGee P, Lund C, Johnson M, Lorenzi G, Gao X, Steffes MW, Lachin JM; GRADE Research Group; DCCT/EDIC Research Group. Comparison of central laboratory HbA1c measurements obtained from a capillary collection versus a standard venous whole blood collection in the GRADE and EDIC studies. PLoS One. 2021 Nov 15;16(11):e0257154. doi: 10.1371/journal.pone.0257154. eCollection 2021. PMID 34780485